CLINICAL TRIAL: NCT03420001
Title: Do Women With Vaginal Birth After Caesarean Section Have an Increased Risk of Levator Avulsion?
Brief Title: Vaginal Birth After Caesarean Section and Levator Ani Avulsion
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Zdenek Rusavy, Principal Investigator, Charles University, Czech Republic
Other Study IDs: 10101010
Record Dates: First submitted 2018-01-27; First posted 2018-02-05 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Birth Injuries
Keywords: VBAC, levator ani avulsion, quality of life
MeSH Terms: conditions — Birth Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VBAC: secundiparous women after one vaginal birth after caesarean section
- controls: women after one vaginal delivery

SUMMARY:
There is no data regarding the risk of levator ani avulsion in women after a vaginal birth after caesarean although a possible increased risk has been suggested. The aim of the study is to describe the incidence of levator ani avulsion and compare it to primiparous women. In addition, health related quality of life will be evaluated and compared

DETAILED DESCRIPTION:
Levator ani muscle avulsion is a frequent postpartum trauma imposing a considerable risk of pelvic organ prolapse on women in later life. Furthermore, the trauma reduces the effectiveness of pelvic reconstructive surgery and has a detrimental effect of the sexuality of the affected women. The trauma occurs most frequently in the first vaginal delivery with an incidence of 10-30%. However, the risk of levator avulsion in women after vaginal birth after caesarean section (VBAC) is unknown although possible increased risk has been suggested.

The aim of the study is to assess the prevalence of levator ani avulsion among women who delivered vaginally after a caesarean section and make a comparison with a primiparous cohort. The secondary aim is to evaluate and compare the health related quality of life regarding pelvic floor disorders and sexuality.

ELIGIBILITY:
Inclusion Criteria:

* one term vaginal delivery in obstetric history
* agreement with the enrollment

Exclusion Criteria:

* Women with a history of repeat VBAC or a vaginal delivery prior to the index caesarean section
* women with preterm labor
* epidural analgesia
* multiple pregnancy
* dead or malformed fetus

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women at least 6 months after the first vaginal delivery with or without a caesarean section in their history.
Sampling Method: Probability Sample
Enrollment: 469 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Levator ani avulsion | at least 6 months after the delivery
  Presence of levator ani avulsion diagnosed by offline tomographic ultrasound imaging of an ultrasound volume of the pelvic floor
Genital hiatus ballooning | at least 6 months after the delivery
  Area of the urogenital hiatus over 25cm2 during maximal Valsalva

SECONDARY OUTCOMES:
Pelvic floor dysfunction | at time of the ultrasound examination
  Pelvic Floor Distress Inventory - PFDI-20 - shortened form of a validated questionnaire evaluating quality of life with pelvic floor disorders (pelvic organ prolapse, urinary incontinence, anal incontinence) evaluation of subscales POPDI-6, UDI-6, CRADI-8 (scale 0-100 in all subscales, the higher the number the higher the impact)
Anal incontinence | at time of the ultrasound examination
  Scoring of the severity of anal incontinence using the St. Mark's score - scoring system (0 - perfect continence, maximum score 24 - totally incontienent.
Sexuality | at time of the ultrasound examination
  Evaluation of sexuality using validated Czech translation of the Pelvic Organ Prolapseand incontinence sexual questionnaire - internationally revised (PISQ-IR) - analysis of individual domains via subscores (NSA-CS, NSA-PR, NSA-GQ, NSA-CI or SA-AO, SA-PR, SA-CS, SA-GQ, SA-D, SA-CI. Transformed score 0-100 for each subscore.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Department of Obstetrics and Gynecology, Medical Faculty in Pilsen, Charles University Hospital, Pilsen
  - Department of Obstetrics and Gynecology, 1st Medical Faculty, Charles University Hospital, Prague

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Horak TA, Guzman-Rojas RA, Shek KL, Dietz HP. Pelvic floor trauma: does the second baby matter? Ultrasound Obstet Gynecol. 2014 Jul;44(1):90-4. doi: 10.1002/uog.13252. Epub 2014 May 23. PMID 24311466
- [Background] Albrich SB, Laterza RM, Skala C, Salvatore S, Koelbl H, Naumann G. Impact of mode of delivery on levator morphology: a prospective observational study with three-dimensional ultrasound early in the postpartum period. BJOG. 2012 Jan;119(1):51-60. doi: 10.1111/j.1471-0528.2011.03152.x. Epub 2011 Oct 10. PMID 21985531
- [Background] Dietz HP, Bernardo MJ, Kirby A, Shek KL. Minimal criteria for the diagnosis of avulsion of the puborectalis muscle by tomographic ultrasound. Int Urogynecol J. 2011 Jun;22(6):699-704. doi: 10.1007/s00192-010-1329-4. Epub 2010 Nov 24. PMID 21107811
- [Background] Dietz HP, Shek C, De Leon J, Steensma AB. Ballooning of the levator hiatus. Ultrasound Obstet Gynecol. 2008 Jun;31(6):676-80. doi: 10.1002/uog.5355. PMID 18470963